CLINICAL TRIAL: NCT01556854
Title: Comparative Effectiveness of Different Neuroprotectants Among Patients With Acute Ischemic Stroke in Clinical Practice
Brief Title: Comparative Effectiveness of Neuroprotectants on Acute Ischemic Stroke
Acronym: CER
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: yongjun wang (Other Government)
Responsible Party: Sponsor-Investigator, yongjun wang, Beijing Tiantan hospital, Ministry of Science and Technology of the People´s Republic of China
Organization: Ministry of Science and Technology of the People´s Republic of China (Other Government)
Other Study IDs: 2011BAI08B02-01
Record Dates: First submitted 2012-03-13; First posted 2012-03-16 (Estimated); Last update posted 2012-03-16 (Estimated); Status verified 2012-03

CONDITIONS: Acute Ischemic Stroke
Keywords: ginkgo leaves; butylphthalide; edaravone; citicoline; cerebrolysin; piracetam; Neuroprotectants
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
The primary objective of this study is to compare effectiveness of five different neuroprotectants, including butylphthalide, edaravone, citicoline, cerebrolysin, and piracetam, among patients with acute ischemic stroke.

The secondary objectives of the study are as follows:

* To compare safety of five different neuroprotectents, including butylphthalide, edaravone, citicoline, cerebrolysin, and piracetam, among patients with acute ischemic stroke.
* To compare cost-effectiveness of five different neuroprotectents, including butylphthalide, edaravone, citicoline, cerebrolysin, and piracetam, among patients with acute ischemic stroke.

DETAILED DESCRIPTION:
Study Population:The study population will consist of consenting patients who are on neuroprotectant injection for the treatment of acute IS during hospitalization. Hospitals may contribute differing numbers of patients to the total sample size. Primary analyses will be conducted on the total sample size only.

Assessment of Outcomes:The outcome measures in this study include effectiveness, safety and cost measures.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old
* Ischemic stroke confirmed by brain CT or MRI within 14 days of the index event
* Neuroprotectents administrated during hospitalization
* Direct admission based on physician evaluation or arrival through the emergency department
* Ability of patient or legally authorized representative (primarily spouse, parents, adult children, otherwise indicated) to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of consenting patients who are on neuroprotectant injection for the treatment of acute IS during hospitalization.
Sampling Method: Probability Sample
Enrollment: 20000 (Estimated)
Dates: Start 2011-07; Primary Completion 2013-11 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
Effectiveness Outcome Measures | 3 years
  * The severity of neurological impairment evaluated by the NIHSS • Disability by mRS
  * All cause mortality
  * In-hospital recurrence and recurrence at 3 month post discharge
  * In-hospital complications
  * Cognitive disorder evaluated by MMSE
  * Quality of Life evaluated by EQ5D

SECONDARY OUTCOMES:
Safety Outcome Measures | 3 years
  * death
  * prolonged inpatient hospitalization
  * a life-threatening experience (that is, immediate risk of dying)
  * persistent or significant disability/incapacity
  * or is considered significant by the physician for any other reason.
Cost-effectiveness Outcome Measures | 2011.7-2014.6
  * Medical cost at discharge
  * Drug cost at discharge
  * Neuroprotectents cost at discharge
  * Administration cost at discharge
  * Medical cost at 3 month post discharge
  * Drug cost at 3 month post discharge

CONTACTS AND LOCATIONS:
Locations (1):
- Tiantan hospital, Beijing, Beijing Municipality, China